CLINICAL TRIAL: NCT01650064
Title: Latin America Hip Fracture Mortality Study
Acronym: LAMOS
Status: Completed | Type: Observational
Sponsor: AO Clinical Investigation and Publishing Documentation (Other)
Responsible Party: Sponsor
Organization: AO Innovation Translation Center (Other)
Other Study IDs: LAMOS
Record Dates: First submitted 2012-07-06; First posted 2012-07-26 (Estimated); Last update posted 2020-08-13 (Actual); Status verified 2017-01

CONDITIONS: Hip Fractures
Keywords: Hip fracture; Mortality
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to estimate the survival proportion one year after surgery for intertrochanteric fracture in older adults in Latin America.

DETAILED DESCRIPTION:
This is a multi-center, prospective, observational clinical study to evaluate mortality in patients with surgically-treated hip fracture in Latin America, and investigate associated prognostic factors. Patients will be followed for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Adults 60 years and older
* Diagnosis of an isolated intertrochanteric fracture (AO 31-A) confirmed by radiographic evaluation
* Primary surgical fracture treatment within 10 days after trauma
* No prior treatment for the fracture
* Ability to understand the content of the patient information / informed consent form
* Willingness and ability to participate in the clinical investigation according to the CIP
* Signed and dated IRB/EC-approved written informed consent

Exclusion Criteria:

* Polytrauma (ie, multiple injuries, whereof one or the combination of several injuries is life threatening)
* Pathologic fracture due to a disease other than osteoporosis (eg, tumor, metastasis)
* Active malignancy
* Class 5 and 6 of the American Society of Anesthesiologists (ASA) physical status classification (Appendix 2)
* Neurological and/or psychiatric disorders that would preclude reliable assessment (eg, Parkinson's disease, multiple sclerosis, severe depression)
* Recent history of substance abuse (ie, recreational drugs, alcohol) that would preclude reliable assessment
* Prisoner
* Participation in any other medical device or medicinal product study within the previous month that could influence the results of the present study
* Noncompletion of patient baseline questionnaires
* Prior implant on the fractured hip

Ages: 60 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with surgically-treated hip fracture in Latin America
Sampling Method: Non-Probability Sample
Enrollment: 168 (Actual)
Dates: Start 2013-01; Primary Completion 2016-04 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Death | after 1 year

SECONDARY OUTCOMES:
Harris Hip Score | Screening/Preoperative and 90 ± 21 days
Parker Mobility Score | Screening/Preoperative, 30±7 days, 60±14 days, 90± 21 days, 365 (up to 425) days
Wound healing | 30±7 days, 60±14 days, and 90± 21 days
Fracture healing | 60±14 days and 90± 21 days
Anticipated surgical treatment-related adverse events | Postoperative (2 to 5 days), 30±7 days, 60±14 days, 90±21 days, 180±121 days, and 365 (up to 425) days
EQ-5D | Screening/Preoperative, 30±7 days, 60±14 days, 90±21 days, 180±121 days, and 365 (up to 425) days

CONTACTS AND LOCATIONS:
Overall Officials: Wiliam Belangero, Dr.med, Principal Investigator — Department of Orthopaedics and Traumatology, Hospital das Clinicas da UNICAMP, Brazil
Locations (16):
- Hospital Italiano de Buenos Aires, Buenos Aires, Argentina
- Brazil (7):
  - Hospital Vila Velha, Espírito Santo
  - IOT - Instituto de Ortopedia de Traumatologia de Passo Fundo, Passo Fundo
  - Hospital Municipal Miguel Couto, Rio de Janeiro
  - Hospital das Clinicas da UNICAMP, São Paulo
  - Hospital Irmandade da Santa Casa de Misericórdia de São Paulo, São Paulo
  - Hospital São Paulo, São Paulo
  - Universidad de São Paulo, São Paulo
- Chile (2):
  - Hospital Clínico Pontificia Universidad Católica de Chile, Santiago
  - Hospital del Trabajador de Santiago, Santiago
- Hospital Infantil de San José, Bogotá, Colombia
- Hospital San Vicente de Paúl, San José, Costa Rica
- Hospital Teodoro Maldonado Carbo, Guayaquil, Ecuador
- Mexico (2):
  - Hospital de Traumatología y Ortopedia "Lomas Verdes", Mexico City
  - Hospital de Traumatología y Ortopedia UMAE #21, Monterrey
- Asociación Española Primera de Socorros Mutuos, Montevideo, Uruguay